CLINICAL TRIAL: NCT04705454
Title: Loncastixumab Tesirine (ADCT-402) Expanded Access Program (EAP) for Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: No longer available | Type: Expanded Access
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADCT-402 EAP
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL)
Keywords: Expanded Access; Lymphoma; Large B-Cell; Relapsed; Refractory
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — loncastuximab tesirine

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Loncastuximab Tesirine
  Other Names: Zynlonta

SUMMARY:
The EAP is for patients with relapsed/refractory diffuse large b-cell lymphoma (R/R DLBCL) that cannot be treated by currently available drugs, cell therapy, or clinical trials. ADC Therapeutics will evaluate patients for approval into the program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 years or older
* Pathologic diagnosis of DLBCL
* Relapsed/Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL) that cannot be treated by currently available drugs, cell therapy, or clinical trials
* Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least six months after the last dose of loncastuximab tesirine. Men with female partners who are of childbearing potential must agree that they will use a highly effective method of contraception from the time of giving informed consent until at least six months after the patient receives his last dose of loncastuximab tesirine

Exclusion Criteria:

* Known history of hypersensitivity to or positive serum human Anti-Drug Antibodies to loncastuximab tesirine
* Total bilirubin >1.5 x upper limit of normal (ULN)
* Active second primary malignancy other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that ADCT Head of Medical Affairs and/or designee, and treating physician agree and document should not be exclusionary
* Autologous Stem Cell Transplantation (SCT) within 30 days prior to start of loncastuximab tesirine
* Allogeneic SCT within 60 days prior to start of loncastuximab tesirine
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
* Lymphoma with active central nervous system involvement at the time of screening, including leptomeningeal disease
* Breastfeeding or pregnant
* Major surgery, radiotherapy, chemotherapy or other anti-neoplastic therapy within 14 days prior to starting loncastuximab tesirine, except shorter if approved by ADCT
* Use of any other experimental medication within 14 days prior to starting loncastuximab tesirine
* Any other significant medical illness, abnormality, or condition that would, in the treating physician's judgment, make the patient inappropriate to receive loncastuximab tesirine or put the patient at risk

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult